CLINICAL TRIAL: NCT00716222
Title: Hormonal and Metabolic Consequences of Sleep Disorders in Young Obese Patients
Acronym: SOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: M.D. PhD V Beauloye, Cliniques universitaires Saint-Luc
Other Study IDs: B40320084032
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Obesity; Sleep Disorders
MeSH Terms: conditions — Obesity; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Obese adolescent and young adult with sleep disorder
- 2: Obese adolescent and young adult without sleep disorder
- 3: Lean adolescent and young adult with sleep disorder

SUMMARY:
There is a well-documented relationship between short sleep duration and high body mass index (BMI). The mechanism linking short sleep duration and weight gain is unknown. Current studies in healthy young volunteers have shown that experimental sleep restriction is associated with dysregulation of the neuroendocrine control of appetite and with alterations in glucose metabolism. The goal of our study is to determine the metabolic and hormonal modifications induced by chronic sleep curtailment in obese adolescents and young adults and to observe if short sleep is a negative prognostic factor in their weight evolution.

DETAILED DESCRIPTION:
The main purpose of the study is investigate whether the concentrations of 2 hormones that regulate appetite (leptin, ghrelin), cytokines (TNF-a, IL-6) and CRP are modified in obese adolescents and young adults who had sleep disorders in comparison to obese adolescents and young adults who sleep longer.

ELIGIBILITY:
Inclusion Criteria:

* 13-25 years old
* BMI > 30 kg/m2 (If adolescents aged under 18 years: BMI equivalent to a BMI for age and sex to a BMI of 30, according to the Cole et al. obesity criteria).

Exclusion Criteria:

* Infection
* Liver disease
* Chronic inflammatory disease
* Endocrine disease
* Use of drugs that alter the sensitivity of insulin

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients of the output clinics in the endocrinology and pediatric endocrinology departments at the university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-05; Study Completion 2009-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Beauloye, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Brussels Capital, Belgium